CLINICAL TRIAL: NCT06868550
Title: Impact of a Comprehensive Oral Health Promotion Program on Maternal Oral Health, Knowledge, Attitudes, and Practices Versus Standard Care in a Group of Egyptian Pregnant Women: a Randomized Controlled Trial
Brief Title: Oral Health Promotion Vs. Standard Care in Egyptian Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Zaki, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CU 26.2.2025
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Maternal and Child Health Outcomes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Behavioral: Comprehensive oral health program: participants will receive structured oral health education through workshops, videos, pamphlets, and interactive support sessions
  Interventions: Behavioral: Comprehensive Oral Health Promotion Program
- Comparator (Active Comparator): Behavioral: Standard oral health care: participants will receive routine oral health education in standard care sessions without additional educational materials or interactive support
  Interventions: Behavioral: Comprehensive Oral Health Promotion Program

INTERVENTIONS:
Behavioral: Comprehensive Oral Health Promotion Program — The principal investigator will carry out all treatment procedures, and the patients will be randomly assigned to any of them.

SUMMARY:
The research question: In pregnant women, does participation in a comprehensive oral health promotion program, compared to standard care, improve maternal oral health, knowledge, attitudes, and practices? This study aims to evaluate the impact of a comprehensive oral health promotion program, compared to standard care, on improving maternal oral health, knowledge, attitudes, and practices among pregnant women. Null hypothesis: There is no significant difference in maternal oral health, knowledge, attitudes, and practices between the group of Egyptian pregnant women who receive the comprehensive oral health promotion program and those who receive standard care. The study population will be pregnant women aged 20 to 45 years. The participants will be categorized into two groups: Intervention will be offered Comprehensive Program and will Include educational workshops, Videos, pamphlets, and support sessions and group chat; and Comparator group will receive Standard care (Limited to oral health sessions only). The study will evaluate three outcomes. Primary outcome The participants will undergo a caries assessment test using The DMFT Index. Secondary outcome The Oral Hygiene Assessment will include the participants using the Simplified Oral Hygiene Index (OHI-S).

Tertiary outcome

1. The knowledge, attitude, and practice (KAP) assessment for pregnant women regarding the Comprehensive Oral Health Promotion Program will be carried out through a prestructured questionnaire. The response data will be collected as frequency and percentage.
2. The nutritional assessment for all participants will be performed using a prestructured questionnaire. The response data will be recorded as frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Mothers willing to participate.
* Pregnant women from 20 to 45 years
* Participants can understand and communicate

Exclusion Criteria:

* Pre-existing systemic conditions such as diabetes or cardiovascular diseases.
* Participants with a high risk of non-compliance with study requirements

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2025-04-12 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Caries assessment | Baseline, 38 weeks
  Participants will undergo a caries assessment test using the Decayed, Missing, and Filled Teeth (DMFT) index. The DMFT index ranges from 0 to 28 (or 32, depending on the number of teeth present). Higher scores indicate worse oral health, as they reflect more decayed, missing, or filled teeth.

SECONDARY OUTCOMES:
Oral Hygiene Assessment | Baseline, Week 12, and week 38
  Participants' oral hygiene status will be assessed using the Simplified Oral Hygiene Index (OHI-S). The OHI-S score ranges from 0 To 6, where higher scores indicate worse oral hygiene due to increased plaque and debris accumlation.

IPD SHARING:
Plan to Share IPD: No
The collected data will not be shared publicly due to confidentiality policies and ethical restrictions.